CLINICAL TRIAL: NCT04664829
Title: Metastatic Triple-Negative Taxane-Resistant Breast Cancer: Investigating the Role of Bexarotene in Inducing Susceptibility to Chemotherapy by Differentiating Cancer Cells From a Mesenchymal-Like to an Epithelial-Like Phenotype
Brief Title: The Role of Bexarotene in Inducing Susceptibility to Chemotherapy in Metastatic TNBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEXMET
Record Dates: First submitted 2020-11-09; First posted 2020-12-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Triple-Negative Breast Carcinoma
Keywords: Bexarotene
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Bexarotene; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bexarotene and Capecitabine (Experimental)
  Interventions: Drug: Bexarotene; Drug: Capecitabine

INTERVENTIONS:
Drug: Bexarotene — Administered orally once a day. Starting dosage: 200mg/m^2
  Other Names: Targretin
Drug: Capecitabine — Administered orally twice a day. Dosage: 1000mg/m^2
  Other Names: Xeloda

SUMMARY:
Triple-negative breast cancer (TNBC) is biologically aggressive and has limited systemic treatment options, often compounded by treatment resistance.

Cell state transitions, e.g. epithelial-to-mesenchymal transition (EMT) govern cancer cell behaviour.

The investigators hypothesize that by inducing change in cell state change, TNBC cells that have manifested taxane-resistance will be more sensitized to subsequent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven metastatic TNBC
* Patients whose TNBC has progressed after prior taxane therapy in the (neo)adjuvant or metastatic setting, and have not received Capecitabine or 5-fluorouracil
* Females aged 21 years and older
* ECOG performance status 0 or 1
* Life expectancy greater than three months
* Patients have normal organ and marrow function
* Site(s) of disease amenable to serial bedside biopsies before, during and after study treatment

Exclusion Criteria:

* Previous palliative radiotherapy to potentially biopsy-able lesion
* Active symptomatic central nervous system (CNS) metastases
* Spinal cord compression not definitively treated with surgery and/or radiation
* Uncontrolled pleural effusion, pericardial effusion, ascites requiring recurrent drainage procedures

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Tumour transcriptome by RNA sequencing | From time of first biopsy before the start of treatment, to disease progression, up to 2 years
  To characterize the changes in tumour transcriptome upon treatment
Tumour protein profile by multiplex immunohistochemistry | From time of first biopsy before the start of study treatment, to disease progression, up to 2 years
  To characterize the changes in tumour protein profile upon treatment

SECONDARY OUTCOMES:
Incidences of treatment related adverse events | From time of start of study treatment, to 28 days after last dose of study treatment, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Lim, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore